CLINICAL TRIAL: NCT06950619
Title: A Clinical Investigation Into the Co-occurrence of Dental Anomalies With Ocular and Cutaneous Features
Brief Title: Associations Between Dental Anomalies and Ocular, Cutaneous and Skin Appendages Features
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pavia (Other)
Responsible Party: Principal Investigator, Andrea Scribante, Associate Professor, Investigator, University of Pavia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2025-DENTALOCULARANOMALIES
Record Dates: First submitted 2025-04-21; First posted 2025-04-30 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Congenital Cataract; Tooth Abnormalities; Ocular Pathologies
MeSH Terms: conditions — Tooth Abnormalities | interventions — Whole Genome Sequencing

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Orthodontic patients (Experimental): Patients fulfilling the inclusion criteria will undergo blood sampling
  Interventions: Genetic: Whole Genome Sequencing; Other: Cephalometric tracing

INTERVENTIONS:
Genetic: Whole Genome Sequencing — Genetic testing will be performed to find variants in genes involving congenital cataract and/or ocular diseases (keratitis, keratoconus, corneal dystrophies, ectopia lentis, glaucoma, retinitis pigmentosa, coloboma and aniridia) and dental anomalies (tooth agenesis, supernumerary teeth, Hutchinson teeth, mulberry molars). Cutaneous appendage anomalies will be also evaluated in clinical history for ascertaining ectodermal diplasia.
Other: Cephalometric tracing — Cephalometric tracing will be performed on lateral cephalometric radiographs if present and not taken on purpose for the study

SUMMARY:
Considering recent literature, it is possible to hypothesise a link between dental anomalies and ocular and/or cutaneous findings, given the existence of shared genetic and developmental mechanisms between these two anatomical areas. Both the eye and teeth develop from ectodermal and mesenchymal tissues, involving common molecular signalling pathways such as Wnt, BMP and PAX. Genetic variants affecting these pathways can therefore determine combined phenotypes, such as congenital cataracts associated with dental agenesis or enamel malformations. Some rare genetic syndromes, such as Nance-Horan syndrome and oculofacio-cardio-dental (OFCD) syndrome, support the hypothesis of a systemic correlation between odontogenesis and ocular development. In a previous study on congenital cataracts, nearly 10% of probands with variants in the BCOR, CWC27, IFIH1, NHS, and PAX6 genes had various dental abnormalities. Therefore, exploring the possible connection between eye and dental diseases may not only facilitate early and multidisciplinary diagnosis, but also open up new perspectives in genetic research and the development of personalised therapeutic approaches, for which whole genome sequencing (WGS) appears to be the first choice for investigating non-syndromic forms. Therefore, the current clinical study aims to identify variants in genes common to eye diseases and dental anomalies (agenesis, supernumerary teeth, Hutchinson's teeth, mulberry molars) in orthodontic patients over the age of 12 with dental anomalies who are about to begin orthodontic treatment or who are attending routine check-ups at the Orthodontics and Paediatric Dentistry Unit, Department of Clinical, Surgical, Diagnostic and Paediatrics Sciences at the University of Pavia who have a family history of ocular and cutaneous manifestations or presenting at the same time dental, ocular and/or cutaneous anomalies. Patients who are eligible will be invited to participate in the study. After signing the informed consent form, the Case Report Form will be completed to collect the data of interest for the study; previous medical reports will be asked to patients or parents/legal guardians in case of minors to ascertain ocular and cutaneous pathologies; a buccal swab will be taken to collect a DNA sample that will be analysed with Next Generation Sequencing. In addition, cephalometric evaluations will be performed if lateral teleradiographs will be available, if already performed in accordance with Good Clinical Practice for the purposes of orthodontic assessment of patients.

ELIGIBILITY:
Inclusion Criteria:

* Supernumerary teeth
* oligodontia
* screw driver sharped incisors
* Hutchinson's teeth
* mulberry molars
* tooth agenesis
* congenital cataract, keratitis, keratoconus, corneal dystrophies, ectopia lentis, glaucoma, retinitis pigmentosa, coloboma and aniridia in probands or relatives
* skin appendages anomalies in probands or relatives

Exclusion Criteria:

* Previous orthodontic, restorative, endodontic, prosthetic and surgical treatment that could alter tooth morphology and position

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Presence of variants in common genes for dental anomalies, ocular diseases and cutaneous/skin appendages features | Baseline
  Whole Genome Sequencing will be used to find pathogenetic variants

SECONDARY OUTCOMES:
SNA angle | Baseline
  Angle between the sella, nasion and A point measured on lateral cephalometric radiograph
SNB angle | Baseline
  Angle between the sella, nasion and B point measured on lateral cephalometric radiograph
ANB angle | Baseline
  Angle between point A, the nasion and point B measured on lateral cephalometric radiograph
SN plane | Baseline
  Plane between the sella point S and nasion point N measured on lateral cephalometric radiograph
ANS-PNS plane | Baseline
  Bispinal plane traced between the anterior nasal spine (ANS) and the posterior nasal spine (PNS) measured on lateral cephalometric radiograph
GoGn plane | Baseline
  Mandibular plane traced between Gonion and Gnathion points measured on lateral cephalometric radiograph
Sella turcica length | Baseline
  Distance between the Tuberculum sellae (TS) and the dorsum sella measured on lateral cephalometric radiograph
Sella turcica diameter | Baseline
  Distance between the Tuberculum Sellae (TS) and the farthest point on the inner wall of the sella measured on lateral cephalometric radiograph
Sella turcica depth | Baseline
  The distance of a line dropped perpendicularly from the interclinoidal distance to the deepest point of the sella floor measured on lateral cephalometric radiograph

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Scribante, Principal Investigator — University of Pavia
Locations (2):
- Italy (2):
  - Unit of Medical Genetics, Department of Molecular Medicine, University of Pavia, Pavia, Lombardy
  - Unit of Orthodontics and Pediatric Dentistry - Section of Dentistry - Department of Clinical, Surgical, Diagnostic and Pediatrics - University of Pavia, Pavia, Lombardy

IPD SHARING:
Plan to Share IPD: No
Data will be available upon motivated request to the Principal Investigator.

REFERENCES:
- [Background] Lecca M, Mauri L, Gana S, Del Longo A, Morelli F, Nicotra R, Plumari M, Galli J, Sirchia F, Valente EM, Cavallari U, Mazza M, Signorini S, Errichiello E. Novel molecular, structural and clinical findings in an Italian cohort of congenital cataract. Clin Genet. 2024 Oct;106(4):403-412. doi: 10.1111/cge.14568. Epub 2024 Jun 5. PMID 38840272